CLINICAL TRIAL: NCT01752686
Title: A Phase III Trial of Carboplatin as Adjuvant Chemotherapy Versus Observation in Triple Negative Breast Cancer With Pathologic Residual Cancer After Neoadjuvant Chemotherapy: POST-Neo Adjuvant Study
Brief Title: A Phase III Trial of Carboplatin as Adjuvant Chemotherapy in Triple Negative Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Byeong Woo Park, Principal Investigator, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Severance_BR_01; DA-TNBC (Other Grant/Funding Number: DA-TNBC)
Record Dates: First submitted 2012-09-26; First posted 2012-12-19 (Estimated); Last update posted 2012-12-25 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: Triple negative breast cancer; adjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- carboplatin chemotherapy (Experimental): At the time of post neo-adjuvant period, the patients will be assigned to each treatment group in a 1:1 ratio i.e. carboplatin AUC 6 group vs. observation group. Six cycles of carboplatin (AUC=6) on the first day of every 21 days.
  Interventions: Drug: carboplatin
- Observation arm (No Intervention): In this observation arm, patients should be follow up with regular interval without treatment.

INTERVENTIONS:
Drug: carboplatin — carboplatin as adjuvant chemotherapy
  Other Names: Adding adjuvant arm
  Arms: carboplatin chemotherapy

SUMMARY:
This study is designed to investigate the efficacy of carboplatin, as a post-operative adjuvant chemotherapy for triple negative breast cancer patients who have pathologic residual cancer after the preoperative chemotherapy.

DETAILED DESCRIPTION:
In Neo-adjuvant period Four cycles of 60 mg/m2 doxorubicin and 600 mg/m2 cyclophosphamide therapy at 3-week intervals followed by four cycles of 100 mg/m2 docetaxel at 3-week intervals.

In POST Neo-adjuvant period

Randomization:

At the time of post neo-adjuvant period, the patients will be assigned to each treatment group in a 1:1 ratio i.e. carboplatin AUC 6 group vs. observation group. Six cycles of carboplatin (AUC=6) on the first day of every 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of breast cancer

  1. Female patients
  2. Histologically confirmed invasive breast cancer

     1. Primary tumor greater than 2cm diameter, measured by mammography and sonography
     2. Any N
  3. ER (estrogen receptor)/ PR (progesterone receptor) / HER2 (negative/ negative/ negative)(ER <1%, PR<1%, IHC 0, 1+ or FISH - in case of IHC (immuno-histochemistry) 2+)
  4. No evidence of metastasis (M0)
  5. No prior hormonal, chemotherapy or radiotherapy is allowed.
  6. No breast operation other than biopsy to make diagnosis is allowed.
  7. Age: 20-years and older, not pregnant pre-, and postmenopausal women with good performance status (ECOG 0-1)
  8. Adequate hematopoietic function: Absolute granulocyte count 1500/mm3, platelet 100,000/mm3, Hemoglobin 10 g/mm3
  9. Adequate renal function: Serum creatinine 1.5 mg/dl
  10. Adequate hepatic function: total bilirubin: 1.5 mg/dl, AST(aspartate aminotransferase)/ALT (alanine transaminase): 2 times normal, Alkaline phosphatase:2 times normal
  11. Written informed consent
  12. Normal mental function to understand and sign the consent
  13. Cardiac function: normal or nonspecific EKG taken within 1 mo of enrollment.
  14. LVEF (left ventricular ejection fraction)50% by MUGA (multiple gated acquisition scan) or Echocardiogram taken within 1 mo of enrollment

Exclusion Criteria:

1. Patients who received hormonal, chemotherapy or radiotherapy for breast cancer
2. Patients who underwent surgery for breast cancer
3. Patients with a history of uncompensated congestive heart failure
4. Patients with inflammatory breast cancer (T4d)
5. Patients without primary tumor (T0)
6. Patients who have history of cancer other than in situ uterine cervix cancer or non-melanotic skin cancer
7. Known hypersensitivity to any of the study drugs

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 587 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | up to 3 years
  To compare DFS between carboplatin and observation within non-pCR (complete remission) patients

SECONDARY OUTCOMES:
overall survival | up to 5years
  To compare overall survival (OS) between carboplatin and observation within non-pCR patients.
pCR rate | up to 3 years
  To assess the pCR rate (no residual invasive carcinoma in primary breast and axillary lymph node) within total TNBC patients.
The percentage of patients who receive breast conserving surgery. | up to 3years
  To assess the percentage of patients who receive breast conserving surgery within total triple negative breast cancer patients
Number of adverse events | up to 3years
  Number of adverse events in patients with non-pCR.

OTHER OUTCOMES:
difference in gene expression pattern | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Byeong Woo Park, MD, PhD, Principal Investigator — Severance Hospital